CLINICAL TRIAL: NCT04590846
Title: The Effectiveness of a Caregiver-mediated Health Educational Intervention on Improving Constipation Among Primary School Children and the Knowledge and Attitude Toward Constipation Among Their Caregivers
Brief Title: A Caregiver-mediated Health Educational Intervention to Improve Constipation Status of Primary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JWang20-JZ01
Record Dates: First submitted 2020-10-11; First posted 2020-10-19 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Constipation
Keywords: constipation; Bristol Stool Scale; health educational intervention
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental design study, which will enroll students in the 3rd to 6th grades of two primary schools and their parents in Yunlin. There will be 200 children in the experimental group and 200 in the control group; with a total of 400 students and their parents. Parents in the experimental group will receive health educational leaflets every week. No intervention will be given to the control group. The 4-weeks intervention is scheduled to be from September to November 2020. Both the experimental and control groups will be asked to fill up a questionnaire at the before and after the intervention. The questionnaire includes the defecation and constipation situation of children, physical activity, dietary behavior, life pressure, and parents' knowledge and attitude toward constipation. Both groups of children have to fill out the Stool diary record sheet once a week, including the intervention period and the follow-up period for a total of 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constipation Health Education (Experimental): Health education leaflets are distributed once a week, and students are asked to bring it back to their parents to read. The activity of "seeing leaflets, accumulating points, and redeeming prizes" is adopted. a reply slip is designed in the weekly health education content, containing 3-5 test questions. Parents need to complete the answers and sign after reading the health education content. Those who have a high degree of correctness and fully paid in within 4 weeks will receive additional points. Students are required to keep a " Stool diary record sheet " every day, and it will be posted in the contact book. Children who have confirmed records and turned in will get 10 points a week, and those who turned in all 8 weeks without random answers can get extra points. The points of the parent health education receipt and the points of the children will be combined and calculated, and the weight will be set according to the total number of points for the draw.
  Interventions: Behavioral: Constipation Health Education Intervention Course; Behavioral: General Health Course
- General Health Course (Active Comparator): In order to correctly evaluate the effectiveness of health education intervention, only the parents of the experimental group will receive the health education leaflet during the intervention period. However, after the end of the trial, an electronic file of parental health education in the control group will be provided. Students are required to keep a " Stool diary record sheet " every day, and it will be posted in the contact book. Children who have confirmed records and turned in will get 10 points a week, and those who turned in all 8 weeks without random answers can get extra points. After the children's points are counted, a lottery will be drawn based on the total number of points. Since the experimental group and the control group have different benchmarks for points, the lottery will be drawn separately from each school. During the lottery process, the time will be announced in advance, and the number will be randomly selected by the computer in a live broadcast method.
  Interventions: Behavioral: General Health Course

INTERVENTIONS:
Behavioral: Constipation Health Education Intervention Course — The 4-weeks health education includes three dimensions. The first is "Causes and Hazards of Constipation". The second is "Constipation Symptoms and Criteria". The third is "Constipation Treatment Strategies and Prevention".
  Health education leaflets with 3 to 5 test questions in the weekly are distributed once a week, students will bring them back to parents, and parents need to complete the answers and sign after reading them.
  Arms: Constipation Health Education
Behavioral: General Health Course — General courses about health issues according to the curriculum of each primary school.

SUMMARY:
The research adopts caregiver-mediated health educational intervention to Improve constipation status of primary school children. It is a quasi-experimental design study, which will enroll students in the 3rd to 6th grades of two primary schools and their parents in Yunlin County. There will be 200 children in the experimental group and 200 in the control group. Parents in the experimental group will receive health educational leaflets every week and no intervention will be given to the control group. Both the experimental and control groups students will be asked to fill up a questionnaire at the before and after the intervention with a total of 8 weeks. The study can provide the understanding of the current status of constipation in primary school children, parents' awareness and attitudes on constipation-related issues.

DETAILED DESCRIPTION:
Background and Purposes: Constipation among children is a global health issue. It can distribute a significant impact on medical, social, and economic dimensions, and can delay children's growth. Without proper treatments on constipation, it would reduce the cure rate and increase recurrence rate. Early diagnosis can improve the prognosis of functional constipation. Only a few studies of children constipation are available in the literature, so it is critical to investigate the topic of constipation among children.

Methods: This is a quasi-experimental design study, which will enroll students in the 3rd to 6th grades of two primary schools and their parents in Yunlin. There will be 200 children in the experimental group and 200 in the control group; a total of 400 students and their parents. Parents in the experimental group will receive health educational leaflets every week and students will have to record the situation of defecation once a week. No intervention will be given to the control group. The 4-weeks intervention is scheduled to be from September to November 2020, with a total of 8 weeks. Both the experimental and control groups will be asked to fill up a questionnaire at the before and after the intervention. The questionnaire includes the defecation and constipation situation of children, physical activity, dietary behavior, life pressure, and parents' knowledge and attitude toward constipation. Both groups of children have to fill out the Stool diary record sheet, including the intervention period and the follow-up period for a total of 8 weeks Children with the first and second types of the Bristol Stool Scale will be defined as constipation.

Expected results: The study can provide the understanding of the current status of constipation in primary school children, parents' awareness and attitudes on constipation-related issues. Besides, through the study, a simple and feasible health educational program for parents of primary school children will be proposed, and the efficacy of the program will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children with grades 3~6 in general classes of primary schools and their primary caregivers

Exclusion Criteria:

* (1) Students who have mild or more server mental disabilities.
* (2) Suspected children with mild cognitive impairment who are receiving resource class services.
* (3) Due to congenital structure, endocrine, small intestinal nerve or muscle abnormalities, abdominal muscle tissue, connective tissue abnormalities, neurological abnormalities, such as irritable bowel syndrome, Hirschsprung disease, milk allergy (lactose intolerance), lupus erythematosus School children in other situations.
* (4) Children with gastrointestinal-related diseases caused by acquired factors such as heavy metals, vitamin D poisoning, drugs, etc.
* (5) School children with intestinal paralysis or slow transmission problems, such as hypothyroidism, hypokalemia, and anal sphincter damage.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The change of parents' knowledge towards constipation related issues between 0-week and 4-week | 0-week, 4-week
  The research tool used in this study is a self-compiled scale of knowledge in the questionnaire. There are 15 items in the scale. For each item, the scoring is 1 or 0 depending on whether a participant's answer is correct or incorrect. Thus the score of this scale ranges from 0 to 15. The higher the score, the better the participant's knowledge of constipation.
The change of parents' attitude towards constipation related issues between 0-week and 4-week | 0-week, 4-week
  The research tool used in this study is a self-compiled scale of attitude in the questionnaire. There are 10 items in the scale. Likert 5-point scale is used for each item, with 1 representing strongly disagree and 5 strongly agree. Thus the score of this scale ranges from 10 to 50. A higher score indicates more positive attitude for constipation improvement and prevention of a participant.
The change of parents' behavior intention towards constipation related issues between 0-week and 4-week | 0-week, 4-week
  The research tool used in this study is a self-compiled scale of behavior intention in the questionnaire. There are 4 items in the scale. Likert 5-point scale is used for each item, with 1 representing strongly disagree and 5 strongly agree. Thus the score of this scale ranges from 4 to 20. A higher score indicates more stronger behavioral intentions for constipation improvement and prevention of a participant.

SECONDARY OUTCOMES:
The numbers of changing constipation status between 0-week and 4-week | 0-week, 4-week
  The numbers of changing constipation status from yes to no and from no to yes between 0-week and 4-week will be recorded and compared.
The numbers of changing constipation status between 0-week and 8-week | 0-week, 8-week
  The numbers of changing constipation status from yes to no and from no to yes between 0-week and 8-week will be recorded and compared.
The incidence rates of constipation at 4-week | 4-week
  Regarding the students without constipation at the baseline (0-week) in the two groups, the incidence rates of constipation in the two groups will be compared after the intervention (4-week).
The incidence rates of constipation at 8-week | 8-week
  Regarding the students without constipation at the baseline (0-week) in the two groups, the incidence rates of constipation in the two groups will be compared at the follow-up time-point (8-week).
The proportions of improved students at 4-week | 4-week
  Regarding the students with constipation at the baseline (0-week) in the two groups, the proportions of students with improved status in the two groups will be compared after the intervention (4-week). Students with constipation at the baseline and becoming free of constipation will be considered "improved".
The proportions of improved students at 8-week | 8-week
  Regarding the students with constipation at the baseline (0-week) in the two groups, the proportions of students with improved status in the two groups will be compared at the follow-up time-point (8-week). Students with constipation at the baseline and becoming free of constipation will be considered "improved".

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Zhen Li, MS, Study Director — Asia University
Locations (2):
- Taiwan (2):
  - Yunlin County Shuicanlin Elementary School, Yuanlin
  - Raoping Elementary School, Yuanlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Axelrod CH, Saps M. The Role of Fiber in the Treatment of Functional Gastrointestinal Disorders in Children. Nutrients. 2018 Nov 3;10(11):1650. doi: 10.3390/nu10111650. PMID 30400292
- [Background] Wu TC, Chen LK, Pan WH, Tang RB, Hwang SJ, Wu L, Eugene James F, Chen PH. Constipation in Taiwan elementary school students: a nationwide survey. J Chin Med Assoc. 2011 Feb;74(2):57-61. doi: 10.1016/j.jcma.2011.01.012. PMID 21354081
- [Background] Yamada M, Sekine M, Tatsuse T. Psychological Stress, Family Environment, and Constipation in Japanese Children: The Toyama Birth Cohort Study. J Epidemiol. 2019 Jun 5;29(6):220-226. doi: 10.2188/jea.JE20180016. Epub 2018 Aug 25. PMID 30146529
- [Result] Asakura K, Masayasu S, Sasaki S. Dietary intake, physical activity, and time management are associated with constipation in preschool children in Japan. Asia Pac J Clin Nutr. 2017 Jan;26(1):118-129. doi: 10.6133/apjcn.112015.02. PMID 28049271